CLINICAL TRIAL: NCT04070768
Title: Phase Ib Study of the Safety and Efficacy of Gemtuzumab Ozogamicin (GO) and Venetoclax in Patients With Relapsed or Refractory CD33+ Acute Myeloid Leukemia:Big Ten Cancer Research Consortium BTCRC-AML17-113
Brief Title: Study of the Safety and Efficacy of Gemtuzumab Ozogamicin (GO) and Venetoclax in Patients With Relapsed or Refractory CD33+ Acute Myeloid Leukemia:Big Ten Cancer Research Consortium BTCRC-AML17-113
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Quigley (Other)
Collaborators: Pfizer (Industry); AbbVie (Industry)
Responsible Party: Sponsor-Investigator, John Quigley, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-AML17-113
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: relapsed; refractory; CD33+
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Gemtuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemtuzumab Ozogamicin(GO) + Venetoclax (Experimental): Gemtuzumab Ozogamicin(GO) + Venetoclax
  Interventions: Drug: Gemtuzumab Ozogamicin; Drug: Venetoclax

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Gemtuzumab Ozogamicin 3mg/m^2, Days 1,4,7
  Other Names: GO
Drug: Venetoclax — Venetoclax, 100,200,400, or 600mg Daily Dose

SUMMARY:
This is a Phase Ib Study to determine the Maximum Tolerated Dose (MTD) of Venetoclax in combination with Gemtuzumab Ozogamicin(GO) in subjects with relapsed/refractory acute myeloid leukemia. Using a standard 3+3 design, subjects will receive once cycle of combination therapy. After one cycle of combination therapy, subjects showing response will continue on to one cycle of consolidation therapy with GO\Veneoclax. Subjects who respond to combination therapy will continue on maintenance Venetoclax until progression or unacceptable toxicity.

Dose-limiting toxicity, defined as an adverse event related (possible, probably, or definite) to Venetoclax and/or Gemtuzumab fulfilling one of the following criteria:

criteria:

* Hematologic toxicity: treatment-related grade 3 or worse neutropenia and/or thrombocytopenia due to bone marrow hypocellularity present at the end of cycle one (day 28) with an additional 28 days allowed for count recovery (i.e. present at day 56); specifically grade 3 or worse neutropenia or thrombocytopenia with the bone marrow documented to be free of leukemic infiltration. Note: patients who enter the study with grade 3 or worse cytopenias will not be evaluable for hematologic dose-limiting toxicities.
* Non-hematologic toxicity: any grade 3 or worse treatment-related toxicity occurring within the first cycle (excluding grade 3-4 infections during cycle one).

The study will also evaluate the Overall Response Rate, Anti-leukemic activity, Relapse-free Survival (RFS), event-free survival (EFS) , and overall survival (OS). The study will evaluate quality of life using the European Organization for the Research and Treatment of Cancer 30 item questionnaire (EORTC QLQ-C30).

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Ages 18 to 75 years at the time of consent.
* ECOG Performance Status of 0-2 within 7 days prior to registration; see Appendix I.
* Patients must have AML, as defined, that is relapsed or refractory. Prior therapy including chemotherapy, immunotherapy, biological or targeted therapy (e.g. FMS-like tyrosine kinase-3 (FLT3) inhibitors, other kinase inhibitors, azacitidine, ATRA) is allowed.
* CD33 expression (by flow or IHC) in at least 20% of the leukemia blasts per local pathologist.
* Prior cancer treatment must be completed at least 21 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤Grade 1 or baseline.
* Demonstrate adequate organ function as defined in the table in the protocol; all screening labs to be obtained within 28 days prior to registration.
* Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Females of childbearing potential and males must be willing to use effective contraception during treatment and for at least 30 days after the last dose of Venetoclax. Females will be advised to use effective contraception for at least 6 months after the last dose of Gemtuzumab and males for at least 3 months after the last dose of Gemtuzumab.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

* Patients with history of prior use of GO or Venetoclax NOTE: Starting with dose cohort 3, prior therapy with venetoclax is allowed, provided patients do not have evidence of p53 deletion or mutations. If the dose cohort is de-escalated to dose cohort 2 due to toxicity in cohort 3, prior exposure to venetoclax will continue to be allowed, provided patients do not have evidence of p53 deletion/mutations.
* History of myeloproliferative neoplasm [MPN] including myelofibrosis, essential thrombocythemia, polycythemia vera, CML with or without BCR-ABL1 translocation, and AML with BCR-ABL1 translocation.
* More than three lines of prior therapy. A line of therapy consists of ≥1 complete cycle of a single agent, a regimen consisting of a combination of several drugs, or a planned sequential therapy of various regimens (e.g., 3-6 cycles of initial therapy with bortezomib-dexamethasone [VD] followed by stem cell transplantation [SCT], consolidation, and lenalidomide maintenance is considered 1 line).
* WBC >25 × 109/L. Cytoreduction is required (hydroxyurea as per local standard of care).
* Acute promyelocytic leukemia.
* Unresolved ≥grade 2 clinically significant nonhematologic toxicities from prior anticancer therapy or unresolved disseminated intravascular coagulation ≥ grade 2 per CTCAE v5 criteria.
* History of other malignancies within 1 year prior to study entry, with the exception of: adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast; basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or treated with other modalities), with curative intent.
* Investigational drug within 4 weeks of study entry.
* History of CHF requiring treatment, left ventricular ejection fraction ≤ 50%, cardiac insufficiency grade III or IV per New York Heart Association classification (NYHA; see Appendix II), or chronic stable angina
* Patients who are HIV positive.
* Known CNS involvement with AML.
* Previous hematopoietic stem cell transplant within 2 months.
* Previous history of veno-occlusive disease/sinusoidal obstruction syndrome.
* Patients who are positive for hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months. Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] may participate.
* Active uncontrolled infection or severe systemic infection. Enrollment is possible after control of infection, at discretion of the treating physician.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Patients who have received strong and/or moderate CYP3A inducers or inhibitors within 7 days prior to the initiation of study treatment unless deemed necessary by the treating physician. (See protocol)
* Patients who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up.
* Unable or unwilling to undergo a screening bone marrow study.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Quigley, MD, Principal Investigator — University of Illinois at Chicago
Locations (4):
- United States (4):
  - Univeristy of Illinois, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2: Gemtuzumab Ozogamicin: Gemtuzumab Ozogamicin 3mg/m^2 IV infusion will be given on days 1,4,7 on cycle 1 and days 1, 4 on cycle 2.
  Venetoclax: Venetoclax 200mg Daily Dose
- Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2: Gemtuzumab Ozogamicin: Gemtuzumab Ozogamicin 3mg/m^2 IV infusion will be given on days 1,4,7 on cycle 1 and days 1, 4 on cycle 2.
  Venetoclax: Venetoclax 400mg Daily Dose
- Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2: Gemtuzumab Ozogamicin: Gemtuzumab Ozogamicin 3mg/m^2 IV infusion will be given on days 1,4,7 on cycle 1 and days 1, 4 on cycle 2.
  Venetoclax: Venetoclax 600mg Daily Dose
Period: Overall Study
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2
Started | 3 | 3 | 12
Completed | 3 | 3 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 12 | 18
Age, Continuous [Median (Full Range); unit: years] | 46 [36 to 63] | 74 [64 to 75] | 60 [22 to 76] | 62 [22 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 5 | 6
  Male | 2 | 3 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 12 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 4
  White | 3 | 3 | 8 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Venetoclax When Administered With Gemtuzumab Ozogamicin (GO)
Description: MTD was determined by testing increasing doses up to 600mg orally daily on dose escalation cohorts 1 to 3 with 3 to 6 participants each. MTD reflects the highest dose of drug where fewer than 33% of subjects experience a dose limiting toxicity (DLT). DLT is defined as an adverse event related (possible, probably, or definite) to Venetoclax and/or Gemtuzumab fulfilling one of the following criteria:
  Hematologic toxicity: treatment-related grade 3 or worse neutropenia and/or thrombocytopenia due to bone marrow hypocellularity present at the end of cycle one (day 28) with an additional 28 days allowed for count recovery (i.e. present at day 56); Note: patients who enter the study with grade 3 or worse cytopenias will not be evaluable for hematologic DLT. Non-hematologic toxicity: any grade 3 or worse treatment-related toxicity occurring within the first 56 days.
Time Frame: 42 days
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint MTD followed a standard "3 + 3" design. Therefore, total participants were 3+3+6=12.
Measure: Number; unit: mg
Groups:
- Gemtuzumab Ozogamicin(GO) + Venetoclax: Gemtuzumab Ozogamicin(GO) + Venetoclax
  Gemtuzumab Ozogamicin: Gemtuzumab Ozogamicin 3mg/m^2, Days 1,4,7
  Venetoclax: Venetoclax, 200,400, or 600mg Daily Dose
Arm/Group | Gemtuzumab Ozogamicin(GO) + Venetoclax
Number analyzed (Participants) | 12
mg | 600

2. Secondary Outcome: Overall Response Rate
Description: Per International Working Group Criteria (IWGC), Complete remission (CR): Bone marrow blasts < 5%; absence of blasts with Auer rods and extramedullary disease; absolute neutrophil count > 1.0 x 109/L(1000/μL); platelet count > 100 x 109/L (100,000/μL); independent of red cell transfusions. CR with incomplete recovery (CRi): All CR criteria except for residual neutropenia < 1.0 x 109/L(1000/μL) or thrombocytopenia < 100 x 109/L (100,000/μL).
  Overall response rate = CR + CRi
Time Frame: Up to 7 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint overall response rate was defined as all patients treated with at least one dose of study drug and have had their disease reevaluated.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 10
Percentage of participants | 0 | 33.3 | 40

3. Secondary Outcome: Anti-leukemic Activity Rate
Description: Per International Working Group Criteria (IWGC), Complete remission (CR): Bone marrow blasts < 5%; absence of blasts with Auer rods and extramedullary disease; absolute neutrophil count > 1.0 x 109/L(1000/μL); platelet count > 100 x 109/L (100,000/μL); independent of red cell transfusions. CR with incomplete recovery (CRi): All CR criteria except for residual neutropenia < 1.0 x 109/L(1000/μL) or thrombocytopenia < 100 x 109/L (100,000/μL). Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
  Anti-leukemic activity Rate =CR+Cri+PR
Time Frame: Up to 7 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Anti-leukemic Activity Rate was defined as all patients treated with at least one dose of study drug and have had their disease reevaluated.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 10
Percentage of participants | 33.3 | 66.7 | 40

4. Secondary Outcome: Relapse-free Survival
Description: Per International Working Group Criteria (IWGC), Complete remission (CR): Bone marrow blasts < 5%; absence of blasts with Auer rods and extramedullary disease; absolute neutrophil count > 1.0 x 109/L(1000/μL); platelet count > 100 x 109/L (100,000/μL); independent of red cell transfusions. CR with incomplete recovery (CRi): All CR criteria except for residual neutropenia < 1.0 x 109/L(1000/μL) or thrombocytopenia < 100 x 109/L (100,000/μL). Relapse: Bone marrow blasts ≥ 5%; or reappearance of blasts in the blood; or development of extramedullary disease.
  Relapse-free survival is defined as the time from achievement of a remission until the relapse or death from any cause in patients achieving CR or CRi. Patients not known to have relapsed or died at last follow-up are censored on the date they were last examined
Time Frame: Up to 7 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Relapse-free survival was defined as all patients treated with at least one dose of study drug and have achieved CR or CRi.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2
Number analyzed (Participants) | 0 | 1 | 4
Months |  | 3.65 [NA to NA] — Not enough events occur to calculate 95% confidence interval. | NA [NA to NA] — Not enough events occur to calculate the median and 95% confidence interval.

5. Secondary Outcome: Event-free Survival
Description: Event-free Survival is defined as the time from on study to treatment failure, disease relapse, or death from any cause. Patients not known to have any of these events are censored on the date of last examined.
Time Frame: 7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 12
Months | 1.08 [1.02 to NA] — Not enough events occur to calculate upper 95% confidence interval. | 3.84 [0.89 to NA] — Not enough events occur to calculate upper 95% confidence interval. | 1.25 [0.95 to NA] — Not enough events occur to calculate upper 95% confidence interval.

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from study entry to death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Time Frame: Up to 8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 12
Months | 6.37 [1.22 to NA] — The analysis is limited to participants who experience failure; there is no censoring. Therefore, the upper 95% confidence interval could not be reached. | 6.11 [5.65 to NA] — The analysis is limited to participants who experience failure; there is no censoring. Therefore, the upper 95% confidence interval could not be reached. | 6.79 [1.84 to NA] — Not enough events occur to calculate upper 95% confidence interval.

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 6/12
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 6/12
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 (N=3) | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 (N=3) | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2 (N=12)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
TUMOR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 4 (5)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Venetoclax 200 mg + Gemtuzumab Ozogamicin 3 mg/m^2 (N=3) | Cohort 2: Venetoclax 400 mg + Gemtuzumab Ozogamicin 3 mg/m^2 (N=3) | Cohort 3: Venetoclax 600 mg + Gemtuzumab Ozogamicin 3 mg/m^2 (N=12)
ANEMIA (Blood and lymphatic system disorders) | 2 (3) | 2 (3) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 2 (2) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (5)
DIARRHEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
EDEMA LIMBS (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 4 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (4)
FEVER (General disorders) | 1 (2) | 1 (1) | 2 (2)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (5)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (8)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
LOCALIZED EDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (7) | 1 (2) | 4 (7)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 2 (3) | 2 (3) | 4 (9)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (3) | 1 (1) | 3 (4)
ANAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (5)
WEIGHT LOSS (Investigations) | 0 (0) | 1 (2) | 1 (2)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
BACTEREMIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
EDEMA FACE (General disorders) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 0 (0) | 0 (0) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
FACIAL PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROPARESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GENERALIZED EDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 0 (0) | 0 (0) | 1 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 4 (5)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
ORAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
THRUSH (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
WEIGHT GAIN (Investigations) | 0 (0) | 0 (0) | 1 (2)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04070768/Prot_SAP_000.pdf